CLINICAL TRIAL: NCT01933789
Title: Health System Intervention to Improve Communication About End-of-Life Care for Vulnerable Patients
Brief Title: Improving Communication About Serious Illness
Acronym: ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, J. Randall Curtis, Professor, Department of Medicine, Division of Pulmonary and Critical Care, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 44023
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Critical Illness; Chronic Disease; Terminal Care; Palliative Care; Communication; Advance Care Planning; Neoplasm Metastasis; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; End Stage Liver Disease; Kidney Failure, Chronic
Keywords: Palliative Care; End-of-Life Issues; Patient/Clinician Communication; Patient/Family Communication; Concordance; Treatment Preferences; Anxiety; Depressive Symptoms; Talking with Your Doctor; Coping with Serious Illness; Outpatient Collaboration
MeSH Terms: conditions — Critical Illness; Chronic Disease; Communication; Neoplasm Metastasis; Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Heart Failure; End Stage Liver Disease; Kidney Failure, Chronic; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Feedback Group (Experimental): Subjects will complete surveys and assessments and will be given the Communication Feedback Form for Patients with Serious Illness to use prior to and during a target outpatient visit.
  Interventions: Behavioral: Communication Feedback Form for Patients with Serious Illness
- Comparison/Usual Care Group (No Intervention): Subjects will only complete surveys and assessments.

INTERVENTIONS:
Behavioral: Communication Feedback Form for Patients with Serious Illness — The intervention, based on self-efficacy theory, identifies patients' preferences for communication about end-of-life care (EOLC) and barriers and facilitators to this communication, and collates these data into a feedback form. The feedback forms are tailored to each recipient (clinician, patient, family) to support the communication tasks which that recipient will address. Feedback forms are sent to participants prior to the target clinic visit. The primary clinician's form suggests referral to palliative care if there are "potentially unmet palliative-care communication needs." All forms include "tips" to help the recipient respond to communication preferences appropriately.
  Other Names: "Audit and Feedback"
  Arms: Feedback Group

SUMMARY:
The purpose of this study is to improve care delivered to patients with serious illness by enhancing communication among patients, families, and clinicians in the outpatient setting. We are testing a new way to help patients share their preferences for talking about end-of-life care with their clinicians and families. To do this we created a simple, short feedback form. The form is designed to help clinicians understand what patients would like to talk about. The goal of this research study is to show that using a feedback form is possible and can be helpful for patients and their families.

DETAILED DESCRIPTION:
Four decades of research on end-of-life care indicate that people who are dying often spend their final days with a significant burden of pain and other symptoms and receive care they would not choose. Patient-clinician communication about end-of-life care is an important focus for improving care for three reasons: 1) when it occurs, it is associated with improved quality of life, reduced anxiety, and fewer intensive life-sustaining therapies at the end of life; 2) physicians frequently do not have discussions about end-of-life care with their patients even though most patients desire these discussions; and 3) our preliminary studies suggest that a simple intervention based on each patient's informational needs and preferences can increase the occurrence and quality of patient-clinician communication about end-of-life care. By tailoring patient-clinician discussions to the individual patient, patients will be able to make care decisions that are best for them and clinicians will be able to provide patients with the care patients' desire.

Our long-term goal is to ensure that patients receive the end-of-life care they desire through improved patient-clinician communication. If effective, this health-system intervention will improve: 1) the occurrence and quality of patient-centered communication about end-of-life care for patients with chronic life-limiting illness and their families; 2) the agreement between patients' wishes for care and care received; and 3) the burden of symptoms of anxiety and depression experienced by patients and families.

We propose a randomized trial of a feedback form, called a "Jumpstart" form, provided to patients, family members and clinicians, specifying the individual patient's communication needs and preferences concerning end-of- life care. The trial will be tested with clinicians (n=120) who provide primary or specialty care to eligible patients at clinics of two large healthcare systems. Eligible patients (up to 6 per clinician, goal n=500) will include those with chronic, life-limiting illness. Family members of patients and interdisciplinary team members of primary clinicians may participate. Primary clinicians will be randomized to the intervention or usual care. The intervention's effectiveness will be compared with usual care using validated self-report questionnaires that will be collected longitudinally (baseline/enrollment, within 2 weeks of the target visit, 3 months, 6 months) from patients and families. Analyses include statistical approaches that take into account that there will be more than one patient for each physician and that data are collected at multiple time points.

Outcomes of this study include patient assessments of: 1) frequency and quality of patient/clinician communication; 2) agreement between care patients desire and care patients receive; and 3) symptoms of anxiety and depression.

We will also use qualitative data to accomplish the following goals: 1) to explore subjects' experiences with the study's activities; 2) to understand barriers to participation; and 3) to explore patient and family experiences with the intervention. To obtain these goals, we will contact a total of 30-40 participants, selected from all subject groups, to participate in one-on-one semi-structured interviews during which they will be asked to share their experiences as a study participant and their perspectives on study activities.

ELIGIBILITY:
Inclusion Criteria:

* Eligible primary clinicians will include all clinicians who provide ongoing primary or specialty care to eligible patient populations. This will include primary care physicians (family medicine and internal medicine), oncologists, pulmonologists, cardiologists, gastroenterologists, nephrologists, neurologists, hepatologists, and geriatricians. Primary clinicians may also include nurse practitioners and physician assistants playing a "primary role" with eligible patients. A "primary role" denotes any clinician for whom having a discussion about end-of-life care with eligible patients would be indicated
* Eligible interprofessional team members will include nurses, social workers and other clinicians who are part of an enrolled primary clinician's clinic team.
* Eligible patients will be those under the care of a participating clinician who are 18 years of age or older, have had 2 or more visits with the primary clinician in the last 18 months, and meet diagnostic criteria. Diagnostic criteria include: 1) metastatic cancer or inoperable lung cancer; 2) chronic obstructive pulmonary disease with FEV1 values <35% predicted or oxygen dependence or restrictive lung disease with a TLC < 50% predicted; 3) New York Heart Association Class III or IV heart failure; 4) Child's Class C cirrhosis or MELD score of >17; 5) dialysis-dependent renal failure and either diabetes or a serum albumin of < 2.5; or, 6) older than 75 years with at least one life-limiting chronic illness or older than 90 years. Additional criteria include: PAH w. 6MWD <250m, restrictive lung disease (IPF, ILD) w/ TLC <50%, and cystic fibrosis with FEV1 < 30%. Eligible patients will also be English-speaking and have no significant dementia or cognitive impairment that would limit his/her ability to complete questionnaires.
* Eligible family members will be identified by the patient, with the criterion that the patient would want the family member involved in medical decision-making for the patient if he/she was not able. For the purpose of this study, "family member" is not confined to legal next-of-kin or immediate family member. Any family member, friend, or caregiver is eligible who is English-speaking and has no dementia or delirium limiting his/her ability to complete questionnaires.

Exclusion Criteria:

* Reasons for exclusion for all subject groups include: legal or risk management concerns; and physical or mental limitations preventing ability to complete research activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Randall Curtis, MD, MPH, Principal Investigator — University of Washington
Locations (6):
- United States (6):
  - Valley Medical Center, Renton, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Northwest Hospital and Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - UW Neighborhood Clinics, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Au DH, Udris EM, Engelberg RA, Diehr PH, Bryson CL, Reinke LF, Curtis JR. A randomized trial to improve communication about end-of-life care among patients with COPD. Chest. 2012 Mar;141(3):726-735. doi: 10.1378/chest.11-0362. Epub 2011 Sep 22. PMID 21940765
- [Background] Knauft E, Nielsen EL, Engelberg RA, Patrick DL, Curtis JR. Barriers and facilitators to end-of-life care communication for patients with COPD. Chest. 2005 Jun;127(6):2188-96. doi: 10.1378/chest.127.6.2188. PMID 15947336
- [Background] Curtis JR, Patrick DL. Barriers to communication about end-of-life care in AIDS patients. J Gen Intern Med. 1997 Dec;12(12):736-41. doi: 10.1046/j.1525-1497.1997.07158.x. PMID 9436892
- [Background] Curtis JR, Engelberg RA, Nielsen EL, Au DH, Patrick DL. Patient-physician communication about end-of-life care for patients with severe COPD. Eur Respir J. 2004 Aug;24(2):200-5. doi: 10.1183/09031936.04.00010104. PMID 15332385
- [Background] Engelberg R, Downey L, Curtis JR. Psychometric characteristics of a quality of communication questionnaire assessing communication about end-of-life care. J Palliat Med. 2006 Oct;9(5):1086-98. doi: 10.1089/jpm.2006.9.1086. PMID 17040146
- [Background] Curtis JR, Wenrich MD, Carline JD, Shannon SE, Ambrozy DM, Ramsey PG. Patients' perspectives on physician skill in end-of-life care: differences between patients with COPD, cancer, and AIDS. Chest. 2002 Jul;122(1):356-62. doi: 10.1378/chest.122.1.356. PMID 12114382
- [Derived] Coats H, Downey L, Sharma RK, Curtis JR, Engelberg RA. Quality of Communication and Trust in Patients With Serious Illness: An Exploratory Study of the Relationships of Race/Ethnicity, Socioeconomic Status, and Religiosity. J Pain Symptom Manage. 2018 Oct;56(4):530-540.e6. doi: 10.1016/j.jpainsymman.2018.07.005. Epub 2018 Jul 17. PMID 30025937
- [Derived] Curtis JR, Downey L, Back AL, Nielsen EL, Paul S, Lahdya AZ, Treece PD, Armstrong P, Peck R, Engelberg RA. Effect of a Patient and Clinician Communication-Priming Intervention on Patient-Reported Goals-of-Care Discussions Between Patients With Serious Illness and Clinicians: A Randomized Clinical Trial. JAMA Intern Med. 2018 Jul 1;178(7):930-940. doi: 10.1001/jamainternmed.2018.2317. PMID 29802770
- [Derived] Fakhri S, Engelberg RA, Downey L, Nielsen EL, Paul S, Lahdya AZ, Treece PD, Curtis JR. Factors Affecting Patients' Preferences for and Actual Discussions About End-of-Life Care. J Pain Symptom Manage. 2016 Sep;52(3):386-94. doi: 10.1016/j.jpainsymman.2016.03.012. Epub 2016 Jun 3. PMID 27265813
- See also: Click here for more information about this study. PCORI Project Summary: Health System Intervention to Improve Communication about End-of-Life Care for Vulnerable Patients — https://www.pcori.org/research-results/2013/health-system-intervention-improve-communication-about-end-life-care
- See also: The End-of-Life Care Research Program at the UW School of Medicine — http://depts.washington.edu/eolcare/
- See also: The Palliative Care Center of Excellence at the University of Washington — http://www.uwpalliativecarecenter.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CLINICIANS and INTERPROFESSIONAL (IP) TEAM recruited from Feb 2014 to Nov 2015. PATIENTS and FAMILY recruited from Mar 2014 to Jun 2016. Potential subjects received introductory letters and phone calls to assess interest and eligibility. INTERVIEWEES were selected via purposive sampling from those who completed the intervention activities.
Pre-assignment Details: 635 CLINICIANS assessed for eligibility; 503 excluded; 132 enrolled. Unit of randomization was clinician. 11 IP TEAM members identified; 4 enrolled. 1113 PATIENTS assessed for eligibility; 576 excluded; 537 enrolled. 142 FAMILY identified; 23 excluded; 119 enrolled. Subjects were enrolled if they completed a baseline survey prior to target visit.
Groups:
- Clinician Intervention; IP Team Intervention; Patient Intervention; Family Member Intervention: Received "Jumpstart" feedback forms and education
- Clinician Control; IP Team Control: Received/Provided usual care, surveys only
- Patient Control; Family Member Control: Received usual care, surveys only
- Interviewees: Key informants: Clinicians, Patients and Family Members
Period: Overall Study
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Started | 65 | 67 | 2 | 2 | 249 | 288 | 58 | 61 | 25
Had Target Visit | 61 (Had target visit(s) completed before clinician or patient withdrawal) | 65 (Had target visit(s) completed before clinician or patient withdrawal) | 2 | 2 | 228 | 266 | 0 | 0 | 0
Completed After-visit Survey | 57 (Number reflects individual clinicians who returned surveys for up to 6 enrolled patients) | 64 (Number reflects individual clinicians who returned surveys for up to 6 enrolled patients) | 2 (Number reflects individual IP Team members who returned surveys for up to 6 enrolled patients) | 1 (Number reflects individual IP Team members who returned surveys for up to 6 enrolled patients) | 0 | 0 | 0 | 0 | 0
Completed 2-Week Survey | 0 | 0 | 0 | 0 | 184 | 215 | 0 | 0 | 0
Completed 3-Month Survey | 0 | 0 | 0 | 0 | 176 | 211 | 37 | 43 | 0
Completed 6-Month Survey | 0 | 0 | 0 | 0 | 160 | 188 | 35 | 40 | 0
Qualitative Interviews | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25
Completed | 59 | 66 | 2 | 1 | 190 | 221 | 43 | 47 | 25
Not Completed | 6 | 1 | 0 | 1 | 59 | 67 | 15 | 14 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 21 | 32 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 8 | 9 | 1 | 4 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 17 | 16 | 1 | 4 | 0
Not completed — Became Ineligible | 4 | 0 | 0 | 0 | 13 | 10 | 13 | 6 | 0

BASELINE CHARACTERISTICS:
Population: Measures do not apply to Interview Subjects (Interviewees). These subjects represent a subset of study participants; interviewees did not separately contribute data and are excluded from the analyses.
Groups:
- Interviewees: Key informants: Clinicians, Patients and Family Members. These subjects did not complete baseline measures.
- Total: Total of all reporting groups
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees | Total
Number analyzed (Participants) | 65 | 67 | 2 | 2 | 249 | 288 | 58 | 61 | 0 | 792
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 65 | 65 | 2 | 2 | 60 | 76 | 28 | 27 |  | 325
  >=65 years | 0 | 2 | 0 | 0 | 189 | 212 | 30 | 34 |  | 467
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (8.64) | 47.2 (10.48) | 41.0 (2.83) | 59.0 (5.66) | 73.6 (11.37) | 73.3 (13.71) | 65.4 (13.32) | 65.3 (13.96) |  | 67.7 (15.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 34 | 2 | 2 | 124 | 132 | 46 | 43 |  | 420
  Male | 28 | 33 | 0 | 0 | 125 | 156 | 12 | 18 |  | 372
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 49 | 51 | 2 | 2 | 206 | 219 | 49 | 51 |  | 629
  Minority Race/Ethnicity | 16 | 16 | 0 | 0 | 43 | 69 | 9 | 8 |  | 161
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 |  | 2
Clinician Type [Count of Participants; unit: Participants] — Binary measure: physician or nurse practicioner Population: Reporting on Clinician subjects only.
  Participants
    number analyzed (Participants) | 65 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 132
    Physician | 60 | 62 |  |  |  |  |  |  |  | 122
    Nurse Practicioner | 5 | 5 |  |  |  |  |  |  |  | 10
Clinician's Specialty [Count of Participants; unit: Participants] — Area of specialization Population: Reporting on Clinician subjects only.
  Participants
    number analyzed (Participants) | 65 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 132
    Family Medicine | 14 | 17 |  |  |  |  |  |  |  | 31
    Internal Medicine | 18 | 18 |  |  |  |  |  |  |  | 36
    Oncology | 8 | 18 |  |  |  |  |  |  |  | 26
    Pulmonology | 3 | 5 |  |  |  |  |  |  |  | 8
    Cardiology | 14 | 3 |  |  |  |  |  |  |  | 17
    Gastroenterology | 3 | 1 |  |  |  |  |  |  |  | 4
    Nephrology | 3 | 4 |  |  |  |  |  |  |  | 7
    Geriatrics | 2 | 1 |  |  |  |  |  |  |  | 3
Competence [Communication & End-of-Life (EOL) Care] [Mean (Standard Deviation); unit: units on a scale] — Clinician self-assessment of competency in talking with patients about end-of-life care using a scale from 1="Not very competent" to 5="Very competent". Population: Questionnaire asked of clinicians at baseline. One intervention clinician did not return a baseline survey.
  units on a scale
    number analyzed (Participants) | 64 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 131
    (all) | 3.8 (0.55) | 3.5 (0.57) |  |  |  |  |  |  |  | 3.8 (0.56)
Patient Self-Assessed Health Status [Median (Inter-Quartile Range); unit: units on a scale] — Five ordinal response options: 0 (excellent), 1 (very good), 2 (good), 3 (fair), 4 (poor) Population: Survey item asked of patients at baseline. Two intervention patients did not provide a valid response.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 247 | 288 | 0 | 0 | 0 | 535
    (all) |  |  |  |  | 2 [2 to 3] | 2 [2 to 3] |  |  |  | 2 [2 to 3]
Patient Education Level [Median (Inter-Quartile Range); unit: units on a scale] — Self-report measure of highest level of education completed: 7 ordinal categories: (0) 8th grade or less, (1) some high school, (2) HS diploma or equivalent, (3) some post-HS education, (4) 4-year college degree, (5) some graduate school, (6) graduate degree. Population: Survey item asked of patients at baseline. One intervention patient did not provide a valid response.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 248 | 288 | 0 | 0 | 0 | 536
    (all) |  |  |  |  | 3 [3 to 4] | 3 [3 to 4] |  |  |  | 3 [3 to 4]
Patient Average Monthly Income [Median (Inter-Quartile Range); unit: units on a scale] — Self-report measure of average pre-tax household monthly income for last 3 years: 8 ordinal categories: (0) no income, (1) $1-$500, (2) $501-$1000, (3) $1001-$1500, (4) $1501-$2000, (5) $2001-$3000, (6) $3001-$4000, (7) $4001 or more. Population: Survey item asked of patients at baseline. Some intervention and control patients did not provide a valid response.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 230 | 270 | 0 | 0 | 0 | 500
    (all) |  |  |  |  | 5 [3 to 7] | 5 [4 to 7] |  |  |  | 5 [3 to 7]
Preference Regarding Future Discussion with Clinician [Count of Participants; unit: Participants] — Patient's indication of desire to avoid future discussion about treatment wishes with the clinician. "Would you like to have a discussion of this type with this doctor?" or "Would you like to have additional discussions with this doctor about this?" Population: Based on survey items asked of patients at baseline.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 249 | 288 | 0 | 0 | 0 | 537
    No objection to future discussion stated |  |  |  |  | 197 | 212 |  |  |  | 409
    Objected to future discussion |  |  |  |  | 52 | 76 |  |  |  | 128
Quality of Communication (QOC): Four-Indicator Latent Construct [Mean (Standard Deviation); unit: scores on a scale] — Quality of Communication: patient ratings of enrolled Clinician on seven aspects of end-of-life communication, each aspect having a pseudo-continuous response range of 0 ('clinician didn't do this') to 11 ('the very best I could imagine').
  Four-Indicator Latent Construct: Measured with QOC items 1, 2, 5, & 6 (measurement invariance imposed between groups and over time) Population: All 4 items answered at baseline & 2 weeks: 127 valid intervention responses; 141 valid control responses.
  Unit of measure: continuous measure with control group mean fixed at zero.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 127 | 141 | 0 | 0 | 0 | 268
    (all) |  |  |  |  | -0.695 (7.089) | 0.000 (6.332) |  |  |  | -0.329 (6.698)
Quality of Communication (QOC): Individual QOC Items [Median (Inter-Quartile Range); unit: units on a scale] — Quality of Communication: patient ratings of clinician on seven aspects of end-of-life communication, each aspect having a pseudo-continuous response range of 0 ('clinician didn't do this') to 11 ('the very best I could imagine').
  Individual QOC Items : all have strong floor effects (resulting in median=0). Population: Survey item asked of patients at baseline. Some intervention and control patients did not provide valid responses on all items.
  units on a scale
    Discuss feelings about getting sicker: number analyzed (Participants) | 0 | 0 | 0 | 0 | 230 | 267 | 0 | 0 | 0 | 497
    Discuss feelings about getting sicker |  |  |  |  | 5.5 [0 to 10] | 8 [0 to 11] |  |  |  | 6 [0 to 11]
    Discuss details about getting sicker: number analyzed (Participants) | 0 | 0 | 0 | 0 | 235 | 266 | 0 | 0 | 0 | 501
    Discuss details about getting sicker |  |  |  |  | 7 [0 to 11] | 8 [0 to 11] |  |  |  | 7 [0 to 11]
    Discuss prognosis: number analyzed (Participants) | 0 | 0 | 0 | 0 | 235 | 273 | 0 | 0 | 0 | 508
    Discuss prognosis |  |  |  |  | 0 [0 to 0] | 0 [0 to 5] |  |  |  | 0 [0 to 0.5]
    Discuss what dying might be like: number analyzed (Participants) | 0 | 0 | 0 | 0 | 239 | 278 | 0 | 0 | 0 | 517
    Discuss what dying might be like |  |  |  |  | 0 [0 to 0] | 0 [0 to 0] |  |  |  | 0 [0 to 0]
    Involve in EOL treatment decisions: number analyzed (Participants) | 0 | 0 | 0 | 0 | 235 | 277 | 0 | 0 | 0 | 512
    Involve in EOL treatment decisions |  |  |  |  | 0 [0 to 8] | 0 [0 to 10] |  |  |  | 0 [0 to 9]
    Ask about important things in life: number analyzed (Participants) | 0 | 0 | 0 | 0 | 237 | 272 | 0 | 0 | 0 | 509
    Ask about important things in life |  |  |  |  | 5 [0 to 11] | 8 [0 to 11] |  |  |  | 6 [0 to 11]
    Ask about spiritual or religious beliefs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 236 | 271 | 0 | 0 | 0 | 507
    Ask about spiritual or religious beliefs |  |  |  |  | 0 [0 to 0] | 0 [0 to 0] |  |  |  | 0 [0 to 0]
Patient Health Questionnaire (PHQ-8): Two-Indicator Latent Construct [Mean (Standard Deviation); unit: scores on a scale] — Patient Health Questionnaire: A self-report measure of depressive symptoms. Eight symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Two-Indicator Latent Construct: Measured with PHQ items 1 & 2 (measurement invariance imposed between groups and over time) Population: Both items answered at baseline, 3-months & 6-months: 117 valid intervention responses; 145 valid control responses.
  Unit of measure: continuous measure with control group mean fixed at zero.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 117 | 145 | 0 | 0 | 0 | 262
    (all) |  |  |  |  | 0.327 (0.706) | 0.000 (0.743) |  |  |  | 0.146 (0.743)
Patient Health Questionnaire (PHQ-8): Eight-Item Scale [Mean (Standard Deviation); unit: scores on a scale] — Patient Health Questionnaire: A self-report measure of depressive symptoms. Eight symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Eight-Item Scale: Sum of responses for the eight symptoms (weighted by 8/7 if only 7 items answered) Population: Survey items asked of patients at baseline. Some intervention and control patients did not provide valid responses on 7+ items.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 245 | 286 | 0 | 0 | 0 | 531
    (all) |  |  |  |  | 5.859 (4.796) | 5.152 (4.744) |  |  |  | 5.478 (4.777)
Generalized Anxiety Disorder (GAD-7): Two-Indicator Latent Construct [Mean (Standard Deviation); unit: scores on a scale] — Generalized Anxiety Disorder: A self-report measure of anxiety symptoms. Seven symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Two-Indicator Latent Construct: Measured with GAD items 1 & 3 (measurement invariance imposed between groups and over time) Population: Both items answered at baseline, 3-months & 6-months: 127 valid intervention responses; 150 valid control responses.
  Unit of measure: continuous measure with control group mean fixed at zero.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 127 | 150 | 0 | 0 | 0 | 277
    (all) |  |  |  |  | 0.179 (0.901) | 0.000 (0.899) |  |  |  | 0.082 (0.903)
Generalized Anxiety Disorder (GAD-7): Seven-Item Scale [Median (Inter-Quartile Range); unit: scores on a scale] — Generalized Anxiety Disorder: A self-report measure of anxiety symptoms. Seven symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Seven-Item Scale: Sum of responses for the seven symptoms (weighted by 7/6 if only 6 items answered). (Strong floor effect) Population: Survey items asked of patients at baseline. Some intervention and control patients did not provide valid responses on 6+ items.
  scores on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 247 | 287 | 0 | 0 | 0 | 534
    (all) |  |  |  |  | 2 [0 to 5] | 1 [0 to 4] |  |  |  | 2 [0 to 4]
Choosing Care [Count of Participants; unit: Participants] — "If you had to make a choice at this time, would you [patient]/your family member [family member] prefer a plan of medical care that focuses on extending your/his or her life as much as possible, even if it means having more pain and discomfort, or would you/he or she want a plan of medical care that focuses on relieving pain and discomfort as much as possible, even if that means not living as long?" Population: Survey items asked of patients & family members at baseline. Two control patients and two control family members did not answer this item.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 249 | 286 | 58 | 59 | 0 | 652
    Extending life |  |  |  |  | 46 | 43 | 12 | 11 |  | 112
    Quality of life (relieving pain and discomfort) |  |  |  |  | 149 | 174 | 32 | 38 |  | 393
    I don't know/Not sure |  |  |  |  | 54 | 69 | 14 | 10 |  | 147
Focus of Care [Count of Participants; unit: Participants] — "Using those same categories, which of the following best describes the focus of the medical care you are currently receiving?" [patient] or "Using those same categories, which of the following best describes the focus of the medical care your family member/friend is currently receiving?" [family member] Population: Survey items asked of patients & family members at baseline. Nine patients [5 intervention and 4 control] and three family members [1 intervention and 2 control] did not answer this item.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 244 | 284 | 57 | 59 | 0 | 644
    Extending life |  |  |  |  | 84 | 113 | 19 | 20 |  | 236
    Quality of life (relieving pain and discomfort) |  |  |  |  | 84 | 90 | 20 | 24 |  | 218
    I don't know/Not sure |  |  |  |  | 76 | 81 | 18 | 15 |  | 190
Barriers [Count of Participants; unit: Participants] — "Which, if any, of the following statements are reasons that you might not want to talk with [your MD/ARNP/PA] about care that you would choose if you were to become very sick?' Answers: Applies to me (true=1) or Does not apply to me (false=0) Population: Survey items asked of patients at baseline. Row values indicate endorsement ("applies to me") of barrier item. Not all patients answered all items.
  Participants
    I don't know what kind of care I would want: number analyzed (Participants) | 0 | 0 | 0 | 0 | 241 | 286 | 0 | 0 | 0 | 527
    I don't know what kind of care I would want |  |  |  |  | 101 | 114 |  |  |  | 215
    I'm not ready to talk about care I would want: number analyzed (Participants) | 0 | 0 | 0 | 0 | 245 | 287 | 0 | 0 | 0 | 532
    I'm not ready to talk about care I would want |  |  |  |  | 55 | 55 |  |  |  | 110
    I don't like to talk about getting very sick: number analyzed (Participants) | 0 | 0 | 0 | 0 | 243 | 288 | 0 | 0 | 0 | 531
    I don't like to talk about getting very sick |  |  |  |  | 69 | 79 |  |  |  | 148
    My doctor never seems to have the time: number analyzed (Participants) | 0 | 0 | 0 | 0 | 237 | 282 | 0 | 0 | 0 | 519
    My doctor never seems to have the time |  |  |  |  | 18 | 25 |  |  |  | 43
    I'd rather concentrate on staying alive: number analyzed (Participants) | 0 | 0 | 0 | 0 | 242 | 285 | 0 | 0 | 0 | 527
    I'd rather concentrate on staying alive |  |  |  |  | 145 | 169 |  |  |  | 314
    I feel that talking about death can bring it close: number analyzed (Participants) | 0 | 0 | 0 | 0 | 241 | 283 | 0 | 0 | 0 | 524
    I feel that talking about death can bring it close |  |  |  |  | 29 | 37 |  |  |  | 66
    I have a living will, so I don't need to talk: number analyzed (Participants) | 0 | 0 | 0 | 0 | 245 | 283 | 0 | 0 | 0 | 528
    I have a living will, so I don't need to talk |  |  |  |  | 51 | 73 |  |  |  | 124
    My ideas about the kind of care I want change: number analyzed (Participants) | 0 | 0 | 0 | 0 | 243 | 285 | 0 | 0 | 0 | 528
    My ideas about the kind of care I want change |  |  |  |  | 107 | 110 |  |  |  | 217
    I have not felt sick enough: number analyzed (Participants) | 0 | 0 | 0 | 0 | 244 | 284 | 0 | 0 | 0 | 528
    I have not felt sick enough |  |  |  |  | 132 | 146 |  |  |  | 278
    I'm not sure which doctor would be caring for me: number analyzed (Participants) | 0 | 0 | 0 | 0 | 242 | 283 | 0 | 0 | 0 | 525
    I'm not sure which doctor would be caring for me |  |  |  |  | 126 | 136 |  |  |  | 262
Facilitators [Count of Participants; unit: Participants] — "People also have a number of reasons for wanting to talk about care that they might choose if they were to become very sick. Which, if any, of the following statements are reasons you might want to discuss care choices with [your MD/ARNP/PA]?' Answers: Applies to me (true) or Does not apply to me (false). Population: Survey items asked of patients at baseline. Row values indicate endorsement ("applies to me") of facilitator item. Not all patients answered all items.
  Participants
    I have been very sick: number analyzed (Participants) | 0 | 0 | 0 | 0 | 243 | 284 | 0 | 0 | 0 | 527
    I have been very sick |  |  |  |  | 130 | 145 |  |  |  | 275
    I have had family or friends who have died: number analyzed (Participants) | 0 | 0 | 0 | 0 | 240 | 285 | 0 | 0 | 0 | 525
    I have had family or friends who have died |  |  |  |  | 161 | 200 |  |  |  | 361
    I worry about the quality of my life in the future: number analyzed (Participants) | 0 | 0 | 0 | 0 | 245 | 285 | 0 | 0 | 0 | 530
    I worry about the quality of my life in the future |  |  |  |  | 132 | 151 |  |  |  | 283
    I worry that I could be a burden: number analyzed (Participants) | 0 | 0 | 0 | 0 | 245 | 285 | 0 | 0 | 0 | 530
    I worry that I could be a burden |  |  |  |  | 171 | 190 |  |  |  | 361

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Discussion About Goals of Care at Target Visit
Description: Patient's response to question, "Did you discuss with this doctor the kind of medical care you would want if you were too sick to speak for yourself?"
Time Frame: 2 weeks after target visit
Population: Patients completing 2-week questionnaires. Not all patients provided data at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 184 | 215 | 0 | 0 | 0
Participants
  Yes |  |  |  |  | 137 | 66 |  |  |
  No or Don't Know |  |  |  |  | 47 | 145 |  |  |
  No response |  |  |  |  | 0 | 4 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p < 0.001, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Bivariate model; there were no confounders; Probit regression coefficient = 1.145, 95% CI 2-sided [0.844 to 1.446] — Control group coded 0; intervention group coded 1

2. Secondary Outcome: Occurrence of Discussion About Goals of Care at Target Visit
Description: Electronic Health Record (EHR) documentation of discussion about advance care planning, prognosis, treatment preference, hospice, palliative care, or Physician Orders for Life-Sustaining Treatment (POLST) at target visit
Time Frame: Target visit
Population: Target visit abstracted from patient electronic health record (EHR); not all data were available for this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  Discussion documented |  |  |  |  | 140 | 45 |  |  |
  Discussion not documented |  |  |  |  | 87 | 220 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p < 0.001, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Bivariate model; there were no confounders; Probit regression coefficient = 1.251, 95% CI 2-sided [0.920 to 1.583] — Control group coded 0; intervention group coded 1

3. Secondary Outcome: Occurrence of Discussion About Goals of Care at Target Visit Among Patients Who Did Not Object to Future Discussion at Baseline
Description: as for outcome 1
Time Frame: 2 weeks after target visit
Population: Patients who completed 2-week questionnaires and reported no objection at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 143 | 164 | 0 | 0 | 0
Participants
  Yes |  |  |  |  | 112 | 44 |  |  |
  No or Don't know |  |  |  |  | 31 | 116 |  |  |
  No response |  |  |  |  | 0 | 4 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p < 0.001, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Bivariate model; there were no confounders; Probit regression coefficient = 1.381, 95% CI 2-sided [1.046 to 1.715] — Control group coded 0; intervention group coded 1

4. Secondary Outcome: Occurrence of Discussion About Goals of Care at Target Visit Among Patients Who Did Not Object to Future Discussion at Baseline
Description: as for outcome 2
Time Frame: Target visit
Population: Patient EHR abstracted for target visit and had no objection at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 180 | 199 | 0 | 0 | 0
Participants
  Discussion documented |  |  |  |  | 114 | 34 |  |  |
  Discussion not documented |  |  |  |  | 66 | 165 |  |  |

5. Secondary Outcome: Goal-Concordant Care
Description: Binary variable indicating whether patient's reported focus of current treatment was concordant with treatment preference
Time Frame: 3 months after target visit
Population: Survey items asked of patients at 3-months. Not all patients provided data at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 176 | 211 | 0 | 0 | 0
Participants
  Discordant |  |  |  |  | 74 | 116 |  |  |
  Concordant |  |  |  |  | 93 | 84 |  |  |
  Unknown (no resp to preference &/or current care) |  |  |  |  | 9 | 11 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Occurrence of goal-concordant care; Test type: Superiority; p = 0.073, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the patient's treatment preference (focus on life extension vs. comfort care); Probit regression coefficient = 0.334, 95% CI 2-sided [-0.031 to 0.699] — Control group coded 0; intervention group coded 1

6. Secondary Outcome: Goal-Concordant Care Among Patients With Stable Treatment Preference
Description: as for outcome 5
Time Frame: 3 months after target visit
Population: Survey items asked of patients at 3-months. Not all patients provided data at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 104 | 103 | 0 | 0 | 0
Participants
  Discordant |  |  |  |  | 27 | 43 |  |  |
  Concordant |  |  |  |  | 74 | 57 |  |  |
  Unknown (no resp to preference &/or current care) |  |  |  |  | 3 | 3 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.017, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; [statistical method as in outcome 5, analysis 1]; Probit regression coefficient = 0.481, 95% CI 2-sided [0.085 to 0.877] — Control group coded 0; intervention group coded 1

7. Secondary Outcome: Quality of Communication (QOC): Four-Indicator Latent Construct
Description: Quality of Communication: patient ratings of clinician on seven aspects of end-of-life communication, each aspect having a pseudo-continuous response range of 0 ('clinician didn't do this') to 11 ('the very best I could imagine').
  Measured with QOC items 1, 2, 5, & 6 (measurement invariance imposed between groups and over time). Outcome is a latent variable, which is not observable, nor is it a composite score that can be mathematically computed (e.g., as a sum or average) from its measured indicators. Instead, it is an abstract construct that is inferred through a mathematical model; it represents a concept and is, therefore, a hypothetical variable.
  Theoretical range: unknown; the latent variable is a hypothetical - not an actual - variable Actual range: inapplicable; cannot be determined; this is an indirectly-measured latent variable; Higher value indicates better outcome (i.e., higher quality communication) Unit of measurement: scores on a scale
Time Frame: 2 weeks from target visit
Population: All 4 items asked of patients at baseline & 2 weeks. Not all patients provided data at these time points.
  Continuous measure with control group mean fixed at zero at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 127 | 141 | 0 | 0 | 0
scores on a scale |  |  |  |  | 4.585 (4.208) | 2.128 (5.570) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.010, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the latent variable as measured at baseline; Probit regression coefficient = 2.022, 95% CI 2-sided [0.476 to 3.569] — Control group coded 0; intervention group coded 1

8. Secondary Outcome: Quality of Communication (QOC): Individual QOC Items
Description: Quality of Communication: patient ratings of clinician on seven aspects of end-of-life communication, each aspect having a pseudo-continuous response range of 0 ('clinician didn't do this') to 11 ('the very best I could imagine').
  Individual QOC Items.
  Theoretical range: 0-11 Actual range: 0-11 Higher value indicates better outcome (i.e., higher quality communication) Unit of measurement: units on a scale
Time Frame: 2 weeks from target visit
Population: Survey items asked of patients at 2-weeks. Not all patients provided data at this time point.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 249 | 288 | 0 | 0 | 0
units on a scale
  Discuss feelings about getting sicker: number analyzed (Participants) | 0 | 0 | 0 | 0 | 172 | 192 | 0 | 0 | 0
  Discuss feelings about getting sicker |  |  |  |  | 10 [6.5 to 11] | 8 [0 to 11] |  |  |
  Discuss details about getting sicker: number analyzed (Participants) | 0 | 0 | 0 | 0 | 169 | 192 | 0 | 0 | 0
  Discuss details about getting sicker |  |  |  |  | 9 [0 to 11] | 8 [0 to 11] |  |  |
  Discuss prognosis: number analyzed (Participants) | 0 | 0 | 0 | 0 | 166 | 193 | 0 | 0 | 0
  Discuss prognosis |  |  |  |  | 0 [0 to 9] | 0 [0 to 9] |  |  |
  Discuss what dying might be like: number analyzed (Participants) | 0 | 0 | 0 | 0 | 165 | 195 | 0 | 0 | 0
  Discuss what dying might be like |  |  |  |  | 0 [0 to 1] | 0 [0 to 0] |  |  |
  Involve in EOL treatment decisions: number analyzed (Participants) | 0 | 0 | 0 | 0 | 165 | 189 | 0 | 0 | 0
  Involve in EOL treatment decisions |  |  |  |  | 9 [0 to 11] | 0 [0 to 10] |  |  |
  Ask about important things in life: number analyzed (Participants) | 0 | 0 | 0 | 0 | 173 | 193 | 0 | 0 | 0
  Ask about important things in life |  |  |  |  | 9 [0 to 11] | 8 [0 to 11] |  |  |
  Ask about spiritual or religion beliefs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 168 | 196 | 0 | 0 | 0
  Ask about spiritual or religion beliefs |  |  |  |  | 0 [0 to 9] | 0 [0 to 4.5] |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about patient's feelings about getting sicker. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p = 0.001, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the outcome variable as measured at baseline; Tobit regression coefficient = 2.209, 95% CI 2-sided [0.939 to 3.479] — Control group coded 0; intervention group coded 1
Statistical Analysis 2: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about details of getting sicker. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p = 0.122, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the outcome variable as measured at baseline; Tobit regression coefficient = 1.237, 95% CI 2-sided [-0.330 to 2.804] — Control group coded 0; intervention group coded 1
Statistical Analysis 3: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about how long the patient might have to live. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p = 0.098, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the outcome variable as measured at baseline and clinician specialty; Tobit regression coefficient = 2.329, 95% CI 2-sided [-0.426 to 5.083] — Control group coded 0; intervention group coded 1
Statistical Analysis 4: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about what dying might be like. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p = 0.352, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Pts clustered under clins. Adjusted for outcome variable as measured at baseline: pt. minority status, education, income; clinician type & specialty; Tobit regression coefficient = 1.573, 95% CI 2-sided [-1.742 to 4.887] — Control group coded 0; intervention group coded 1
Statistical Analysis 5: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about patient's involvement in end-of-life treatment decisions. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p < 0.001, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the outcome variable as measured at baseline; Tobit regression coefficient = 4.625, 95% CI 2-sided [2.060 to 7.190] — Control group coded 0; intervention group coded 1
Statistical Analysis 6: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about things in life that are important to the patient. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p = 0.002, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the outcome variable as measured at baseline; Tobit regression coefficient = 2.404, 95% CI 2-sided [0.898 to 3.909] — Control group coded 0; intervention group coded 1
Statistical Analysis 7: Comparison: Patient Intervention vs Patient Control; Patient rating of clinician's quality of communication about patient's religious/spiritual beliefs. Variable with range 0-11, defined as censored from below because of strong floor effect; Test type: Superiority; p = 0.075, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for the outcome variable as measured at baseline and clinician type; Tobit regression coefficient = 2.455, 95% CI 2-sided [-0.250 to 5.159] — Control group coded 0; intervention group coded 1

9. Secondary Outcome: Patient Health Questionnaire (PHQ-8): Two-Indicator Latent Construct
Description: Patient Health Questionnaire: A self-report measure of depressive symptoms. Eight symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Two-Indicator Latent Construct: Measured with PHQ items 1 & 2 (measurement invariance imposed between groups and over time). Outcome is a latent variable, which is not observable, nor is it a composite score that can be mathematically computed (e.g., as a sum or average) from its measured indicators. Instead, it is an abstract construct that is inferred through a mathematical model; it represents a concept and is, therefore, a hypothetical variable.
  Theoretical range: unknown; the latent variable is a hypothetical - not an actual - variable Actual range: inapplicable; cannot be determined; this is an indirectly-measured latent variable Higher value indicates worse outcome (i.e., higher level of depressive symptoms) Unit of measurement: scores on a scale
Time Frame: 3 months after target visit
Population: Both survey items answered by patients at baseline, 3-months & 6-months: 117 valid intervention responses; 145 valid control responses.
  Continuous measure with control group mean fixed at zero.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 117 | 145 | 0 | 0 | 0
scores on a scale |  |  |  |  | 0.255 (0.804) | 0.199 (0.722) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of depression - Two-indicator latent variable with measurement invariance imposed between groups and over time; Test type: Superiority; p = 0.369, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for baseline level of the latent depression variable and for the patient racial/ethnic minority status; Probit regression coefficient = -0.103, 95% CI 2-sided [-0.327 to 0.122] — Control group coded 0; intervention group coded 1

10. Secondary Outcome: Patient Health Questionnaire (PHQ-8): Eight-Item Scale
Description: Patient Health Questionnaire: A self-report measure of depressive symptoms. Eight symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Eight-Item Scale: Sum of responses for the eight symptoms (weighted by 8/7 if only 7 items answered).
  Theoretical range: 0-24 Actual range: 0-24 Higher value indicates worse outcome (i.e., higher level of depressive symptoms) Unit of measurement: scores on a scale
Time Frame: 3 months after target visit
Population: Survey items asked of patients at baseline. Some intervention and control patients did not provide valid responses on 7+ items.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 167 | 195 | 0 | 0 | 0
scores on a scale |  |  |  |  | 5.879 (4.776) | 4.908 (4.634) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of depression: standard PHQ-8 composite score; Test type: Superiority; p = 0.536, Clustered robust linear regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for baseline level of the PHQ-8 composite score; Probit regression coefficient = 0.263, 95% CI 2-sided [-0.571 to 1.097] — Control group coded 0; intervention group coded 1

11. Secondary Outcome: Patient Health Questionnaire (PHQ-8): Two-Indicator Latent Construct
Description: as for outcome 9
Time Frame: 6 months after target visit
Population: Both survey items answered by patients at baseline, 3-months & 6-months: 117 valid intervention responses; 145 valid control responses.
  Continuous measure with control group mean fixed at zero at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 117 | 145 | 0 | 0 | 0
scores on a scale |  |  |  |  | 0.399 (0.873) | 0.244 (0.737) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of depression: Two-indicator latent variable with measurement invariance imposed between groups and over time; Test type: Superiority; p = 0.106, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Pts clustered under clins. Adjusted for baseline level of the latent depression var; pt age, minority status, education, health status; clin specialty; Probit regression coefficient = 0.208, 95% CI 2-sided [-0.044 to 0.461] — Control group coded 0; intervention group coded 1

12. Secondary Outcome: Patient Health Questionnaire (PHQ-8): Eight-Item Scale
Description: as for outcome 10
Time Frame: 6 months after target visit
Population: Survey items asked of patients at 6-months. Some intervention and control patients did not provide valid responses on 7+ items.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 146 | 171 | 0 | 0 | 0
scores on a scale |  |  |  |  | 5.853 (5.339) | 4.850 (4.410) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of depression: Standard PHQ-8 composite score; Test type: Superiority; p = 0.343, Clustered robust linear regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for baseline level of the PHQ-8 composite score and clinician specialty; Probit regression coefficient = 0.446, 95% CI 2-sided [-0.476 to 1.368] — Control group coded 0; intervention group coded 1

13. Secondary Outcome: Generalized Anxiety Disorder (GAD-7): Two-Indicator Latent Construct
Description: Generalized Anxiety Disorder: A self-report measure of anxiety symptoms. Seven symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Two-Indicator Latent Construct: Measured with GAD items 1 & 2 (measurement invariance imposed between groups and over time). Outcome is a latent variable, which is not observable, nor is it a composite score that can be mathematically computed (e.g., as a sum or average) from its measured indicators. Instead, it is an abstract construct that is inferred through a mathematical model; it represents a concept and is, therefore, a hypothetical variable.
  Theoretical range: unknown; the latent variable is a hypothetical - not an actual - variable Actual range: inapplicable; cannot be determined; this is an indirectly-measured latent variable Higher value indicates worse outcome (i.e., higher level of anxiety symptoms) Unit of measurement: scores on a scale
Time Frame: 3 months after target visit
Population: Both survey items answered by patients at baseline, 3-months & 6-months: 127 valid intervention responses; 150 valid control responses.
  Continuous measure with control group mean fixed at zero at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 127 | 150 | 0 | 0 | 0
scores on a scale |  |  |  |  | 0.281 (0.788) | 0.217 (0.807) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of anxiety: Two-indicator latent variable with measurement invariance imposed between groups and over time; Test type: Superiority; p = 0.734, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for baseline level of the latent anxiety variable; Probit regression coefficient = -0.034, 95% CI 2-sided [-0.232 to 0.163] — Control group coded 0; intervention group coded 1

14. Secondary Outcome: Generalized Anxiety Disorder (GAD-7): Seven-Item Scale
Description: Generalized Anxiety Disorder: A self-report measure of anxiety symptoms. Seven symptoms, each with ordinal response options, each option associated with a text description ranging from 'Not at all' to 'Nearly every day'.
  Seven-Item Scale: Sum of responses for the seven symptoms (weighted by 7/6 if only 6 items answered). (Strong floor effect.)
  Theoretical range: 0-21 Actual range: 0-21 Higher value indicates worse outcome (i.e., higher level of anxiety symptoms) Unit of measurement: scores on a scale
Time Frame: 3 months after target visit
Population: Survey items asked of patients at 3-months. Some intervention and control patients did not provide valid responses on 6+ items.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 171 | 196 | 0 | 0 | 0
scores on a scale |  |  |  |  | 2 [0 to 5] | 2 [0 to 4] |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of anxiety: Standard GAD-7 composite score; Test type: Superiority; p = 0.935, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Pts clustered under clins. Clustered Tobit regression because strong floor effect on composite score. Adjusted for baseline level of composite score; Tobit regression coefficient = 0.041, 95% CI 2-sided [-0.946 to 1.028] — Control group coded 0; intervention group coded 1

15. Secondary Outcome: Generalized Anxiety Disorder (GAD-7): Two-Indicator Latent Construct
Description: as for outcome 13
Time Frame: 6 months after target visit
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 127 | 150 | 0 | 0 | 0
scores on a scale |  |  |  |  | 0.297 (0.847) | 0.209 (0.935) |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Symptoms of anxiety: Two-indicator latent variable with measurement invariance imposed between groups and over time; Test type: Superiority; p = 0.689, Clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance; Patients clustered under clinicians. Adjusted for baseline level of the latent anxiety variable; Probit regression coefficient = -0.042, 95% CI 2-sided [-0.247 to 0.163] — Control group coded 0; intervention group coded 1

16. Secondary Outcome: Generalized Anxiety Disorder (GAD-7): Seven-Item Scale
Description: as for outcome 14
Time Frame: 6 months after target visit
Population: Survey items asked of patients at 6-months. Some intervention and control patients did not provide valid responses on 6+ items.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 153 | 176 | 0 | 0 | 0
scores on a scale |  |  |  |  | 1 [0 to 6] | 1 [0 to 4] |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.852, Clustered Tobit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance. Patients clustered under clinicians. Clustered Tobit regression because of strong floor effect on composite score; Adjusted for baseline level of the GAD-7 composite score; Tobit regression coefficient = -0.105, 95% CI 2-sided [-1.204 to 0.995] — Control group coded 0; intervention group coded 1

17. Secondary Outcome: Avoidance of Life-Sustaining Therapies, All Patients
Description: Review of EHR documentation to assess use of three indicators of life-sustaining therapies (LST): admission to an ICU, receipt of CPR, and receipt of mechanical ventilation
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  Received LST |  |  |  |  | 18 | 14 |  |  |
  Avoided LST |  |  |  |  | 209 | 251 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.418, clustered probit regression — No adjustment for multiple tests. A priori threshold of 0.05 for statistical significance. Patients clustered under clinicians; Adjusted for confounding by patient race and health status and by clinician type and specialty; probit regression coefficient = -0.221, 95% CI 2-sided [-0.923 to 0.482] — Control group coded 0; intervention group coded 1

18. Secondary Outcome: Avoidance of Life-Sustaining Therapies, Patients With Comfort Care Preference
Description: Review of EHR documentation to assess use of three indicators of life-sustaining therapies (LST): admission to an ICU, receipt of CPR, and receipt of mechanical ventilation for patients preferring "comfort" (quality of life over extending life) at the end-of-life
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 109 | 112 | 0 | 0 | 0
Participants
  Received LST |  |  |  |  | 7 | 10 |  |  |
  Avoided LST |  |  |  |  | 102 | 102 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.568, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = 0.175, 95% CI 2-sided [-0.613 to 0.962] — Control group coded 0; intervention group coded 1

19. Secondary Outcome: Palliative Care Consultation, Inpatient Stay - All Patients
Description: EHR documentation of palliative care consultation during an inpatient stay for all patients with target visit and chart abstraction.
Time Frame: 3-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  No |  |  |  |  | 221 | 260 |  |  |
  Yes |  |  |  |  | 6 | 5 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.592, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = 0.140, 95% CI 2-sided [-0.534 to 0.815] — Control group coded 0; intervention group coded 1

20. Other Pre Specified Outcome: Group Differences - Treatment Preference (Adjustment Variable for Outcome Measuring Goal-concordant Care)
Description: Binary variable indicating whether patient's current preference was for life-extension or comfort care
Time Frame: 3 months after target visit
Population: Patients completing 3-month questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 176 | 211 | 0 | 0 | 0
Participants
  Life extension |  |  |  |  | 33 | 31 |  |  |
  Comfort |  |  |  |  | 104 | 121 |  |  |
  Unsure |  |  |  |  | 34 | 52 |  |  |
  No response |  |  |  |  | 5 | 7 |  |  |

21. Other Pre Specified Outcome: Group Differences - Stable Treatment Preference (Filter for Subgroup Analysis of Goal-concordant Care)
Description: Binary variable indicating whether patient's treatment preference was stable between target visit (or baseline, if no 2-week questionnaire was returned) and 3 months.
Time Frame: 3 months after target visit
Population: Patients completing 3-month questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 176 | 211 | 0 | 0 | 0
Participants
  Stable |  |  |  |  | 104 | 103 |  |  |
  Not stable |  |  |  |  | 12 | 13 |  |  |
  Unknown (pref not stated at one or both time pts) |  |  |  |  | 60 | 95 |  |  |

22. Secondary Outcome: Palliative Care Consultation, Inpatient Stay - Patients Most Likely to Benefit
Description: EHR documentation of palliative care consultation during an inpatient stay for patients who reported preference for "comfort care" (quality of life over extending life) and wanted a discussion.
Time Frame: 3-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 87 | 110 | 0 | 0 | 0
Participants
  No |  |  |  |  | 86 | 102 |  |  |
  Yes |  |  |  |  | 1 | 8 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.705, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.179, 95% CI 2-sided [-1.398 to 1.040] — Control group coded 0; intervention group coded 1

23. Secondary Outcome: Palliative Care Consultation, Inpatient Stay - All Patients
Description: as for outcome 19
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  No |  |  |  |  | 218 | 257 |  |  |
  Yes |  |  |  |  | 9 | 8 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.644, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = 0.123, 95% CI 2-sided [-0.560 to 0.805] — Control group coded 0; intervention group coded 1

24. Secondary Outcome: Palliative Care Consultation, Inpatient Stay - Patients Most Likely to Benefit
Description: as for outcome 22
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 93 | 119 | 0 | 0 | 0
Participants
  No |  |  |  |  | 91 | 114 |  |  |
  Yes |  |  |  |  | 2 | 5 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.908, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; Adjusted for confounding by patient education and health status and by clinician gender; probit regression coefficient = -0.165, 95% CI 2-sided [-3.833 to 3.503] — Control group coded 0; intervention group coded 1

25. Secondary Outcome: Palliative Care Referral, Outpatient Visit - All Patients
Description: EHR documentation of referral to palliative care services, or discussion about a referral, during an outpatient visit.
Time Frame: 3-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  No |  |  |  |  | 217 | 250 |  |  |
  Yes |  |  |  |  | 10 | 15 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.552, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.121, 95% CI 2-sided [-0.646 to 0.403] — Control group coded 0; intervention group coded 1

26. Secondary Outcome: Palliative Care Referral, Outpatient Visit - Patients Most Likely to Benefit
Description: EHR documentation of referral to palliative care services, or discussion about a referral, during an outpatient visit for patients who reported preference for "comfort care" (quality of life over extending life) and wanted a discussion.
Time Frame: 3-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 87 | 110 | 0 | 0 | 0
Participants
  No |  |  |  |  | 84 | 103 |  |  |
  Yes |  |  |  |  | 3 | 7 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.372, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.293, 95% CI 2-sided [-1.139 to 0.553] — Control group coded 0; intervention group coded 1

27. Secondary Outcome: Palliative Care Referral, Outpatient Visit - All Patients
Description: EHR documentation of referral to palliative care services, or discussion about a referral, during an outpatient visit.
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  No |  |  |  |  | 213 | 244 |  |  |
  Yes |  |  |  |  | 14 | 21 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.501, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.130, 95% CI 2-sided [-0.630 to 0.369] — Control group coded 0; intervention group coded 1

28. Secondary Outcome: Palliative Care Referral, Outpatient Visit - Patients Most Likely to Benefit
Description: as for outcome 26
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 93 | 119 | 0 | 0 | 0
Participants
  No |  |  |  |  | 89 | 108 |  |  |
  Yes |  |  |  |  | 4 | 11 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.192, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.390, 95% CI 2-sided [-1.160 to 0.380] — Control group coded 0; intervention group coded 1

29. Secondary Outcome: Palliative Care Consultation and/or Referral - All Patients
Description: EHR documentation of palliative care referral during an outpatient visit and/or palliative care consultation during an inpatient stay.
Time Frame: 3-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  No |  |  |  |  | 212 | 247 |  |  |
  Yes |  |  |  |  | 15 | 18 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.940, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.014, 95% CI 2-sided [-0.489 to 0.461] — Control group coded 0; intervention group coded 1

30. Secondary Outcome: Palliative Care Consultation and/or Referral - Patients Most Likely to Benefit
Description: EHR documentation of palliative care referral during an outpatient visit and/or palliative care consultation during an inpatient stay for patients who reported preference for "comfort care" (quality of life over extending life) and wanted a discussion.
Time Frame: 3-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 87 | 110 | 0 | 0 | 0
Participants
  No |  |  |  |  | 83 | 102 |  |  |
  Yes |  |  |  |  | 4 | 8 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.470, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.229, 95% CI 2-sided [-1.044 to 0.587] — Control group coded 0; intervention group coded 1

31. Secondary Outcome: Palliative Care Consultation and/or Referral - All Patients
Description: as for outcome 29
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 227 | 265 | 0 | 0 | 0
Participants
  No |  |  |  |  | 206 | 240 |  |  |
  Yes |  |  |  |  | 21 | 25 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.955, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.010, 95% CI 2-sided [-0.474 to 0.454] — Control group coded 0; intervention group coded 1

32. Secondary Outcome: Palliative Care Consultation and/or Referral - Patients Most Likely to Benefit
Description: as for outcome 30
Time Frame: 6-month period following the target visit
Population: Patients who had a target visit and a chart reviewed.
Measure: Count of Participants; unit: Participants
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 93 | 119 | 0 | 0 | 0
Participants
  No |  |  |  |  | 87 | 106 |  |  |
  Yes |  |  |  |  | 6 | 13 |  |  |
Statistical Analysis 1: Comparison: Patient Intervention vs Patient Control; Test type: Superiority; p = 0.303, clustered probit regression — [p-value comment as in outcome 17, analysis 1]; No covariate adjustment; probit regression coefficient = -0.287, 95% CI 2-sided [-1.005 to 0.431] — Control group coded 0; intervention group coded 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study activities: 42 months.
Arm/Group | Clinician Intervention | Clinician Control | IP Team Intervention | IP Team Control | Patient Intervention | Patient Control | Family Member Intervention | Family Member Control | Interviewees
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/67 | 0/2 | 0/2 | 0/249 | 0/288 | 0/58 | 0/61 | 0/25
Other Adverse Events (participants affected / at risk) | 0/65 | 0/67 | 0/2 | 0/2 | 0/249 | 2/288 | 0/58 | 0/61 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clinician Intervention (N=65) | Clinician Control (N=67) | IP Team Intervention (N=2) | IP Team Control (N=2) | Patient Intervention (N=249) | Patient Control (N=288) | Family Member Intervention (N=58) | Family Member Control (N=61) | Interviewees (N=25)
Subject complaint (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Complaint and/or concerns with end-of-life / palliative care aspects of survey

LIMITATIONS AND CAVEATS:
This study took place in one region of the US and may not generalize to other regions. There may be selection bias among those clinicians and patients who were willing to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No